CLINICAL TRIAL: NCT05680766
Title: Feasibility Assessment of Cardiovascular Endurance Training for the Symptomatic Improvement of Irritable Bowel Syndrome Patients With a Sedentary and Non-active Lifestyle.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Face-IT
Record Dates: First submitted 2022-12-23; First posted 2023-01-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: IBS subjects fulfilling the eligibility criteria will follow a structured and personalised cardiovascular endurance training (CET).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): IBS subjects fulfilling the eligibility criteria will follow a structured and personalised cardiovascular endurance training (CET).
  Interventions: Other: Cardiovascular endurance training

INTERVENTIONS:
Other: Cardiovascular endurance training — Based on the results of a maximal effort test, investigators will provide a personalised training program. Results of a submaximal effort test after 6 weeks, will allow for adaptation of the training program for the remaining training period.

SUMMARY:
This exploratory study's primary objective is the changes of irritable bowel syndrome (IBS) symptom severity by cardiovascular endurance training (CET) in relation to the baseline sedentary or non-active lifestyle. Secondary endpoints focus on the mechanisms associated with these changes.

These mechanisms relate to dietary adaptations, changes in anxiety, depressive comorbidity, somatisation, alterations in the gut microbiome or metabolome, body composition and measures of cardiovascular fitness. Virtually all IBS guidelines mention lifestyle modifications as a management option.

Research on the role of physical activity remains underassessed as compared to the other interventions. Therefore, an exploratory proof-of-concept study will investigate the influence of regular physical exercise on symptoms in a small group of IBS patients. This study will gather data on putative underlying mechanisms related to dietary factors, faecal microbiome and metabolome, mental well-being, body composition and cardiovascular fitness.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 60 years;
* Fulfilling the ROME IV criteria for Irritable bowel syndrome (IBS);
* Moderate symptom severity as defined by a IBS-Symptom Severity Scale > 175;
* Sedentary lifestyle defined as SIT-Q-7D > 8h/day;
* Physically inactive defined as < 150min/week on the IPAQ score

Exclusion Criteria:

* Cardiorespiratory disorder hampering participation in a program of physical exercise as evidenced by the sport + keuringsartsen (SKA) questionnaire.
* Clinical suspicion of an organic disorder different from IBS (patients can be included when this disorder had been excluded);
* Known inflammatory bowel disorder;
* Known intestinal motility disorder;
* Alcohol (defined as more than 14 U per week) or other substance abuse;
* Active psychiatric disorder;
* Known systemic or auto-immune disorder with implication for the GI system;
* Prior abdominal surgery (with the exception of appendectomy or cholecystectomy more than 6 months ago);
* Any prior diagnosis of cancer other than basocellular carcinoma;
* Current chemotherapy;
* History of gastro-enteritis in the past 8 weeks;
* Change in diet in the past 8 weeks;
* Dietary supplements unless taken at a stable dose for more than 8 weeks;
* Antibiotics, pre-, pro-, post-biotics or any combination during the past 8 weeks;
* Treatment with neuromodulators (one neuromodulator taken at a stable dose for more than 12 weeks is allowed);
* Treatment with spasmolytic agents, opioids, loperamide, gelatine tannate or mucoprotect-ants during the past 8 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-01-02 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Change of IBS Symptom severity | from baseline to 12 weeks
  this will be assessed after patients have done a cardiovascular endurance training

SECONDARY OUTCOMES:
Change of IBS Symptom severity | from baseline to 6 weeks
  this will be assessed after patients have done a cardiovascular endurance training

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: Undecided